CLINICAL TRIAL: NCT01661595
Title: The Effect of Sildenafil and Tadalafil on Skeletal Muscle and Perceptual Fatigue.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-153
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-04

CONDITIONS: Fatigue
Keywords: Fatigue; Fatigability; Surface Electromyography (sEMG); cyclic guanosine monophosphate (cGMP); Nitric Oxide (NO); NO-cGMP; Phosphodiesterase (PDE); Sildenafil; Tadalafil; Isotope; Infusion; Anabolism; Upregulation; Accelerometer; Placebo; Nitrosylation
MeSH Terms: conditions — Fatigue | interventions — Sildenafil Citrate; Tadalafil

STUDY DESIGN:
Intervention Model Description: Subjects were assigned to one of 4 arms:
  1. Sildenafil (50mg/day) for weeks 0-4. Placebo for weeks 5-8.
  2. Tadalafil (10mg/day) for weeks 0-4. Placebo for weeks 5-8.
  3. Placebo for weeks 0-4. Sildenafil (50mg/day) for weeks 5-8.
  4. Placebo for weeks 0-4. Tadalafil (10mg/day) for weeks 5-8.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sildenafil / Placebo (Active Comparator): 50 mg/day Sildenafil: (Other Name: Viagra, Revatio) for weeks 0-4. Placebo for weeks 5-8.
  Interventions: Drug: Sildenafil; Drug: Placebo
- Tadalafil / Placebo (Active Comparator): 10 mg/day Tadalafil: (Other Name: Cialis, Adcirca) for weeks 0-4. Placebo for weeks 5-8.
  Interventions: Drug: tadalafil; Drug: Placebo
- Placebo / Sildenafil (Active Comparator): Placebo for weeks 0-4. 50 mg/day Sildenafil: (Other Name: Viagra, Revatio) for weeks 5-8.
  Interventions: Drug: Sildenafil; Drug: Placebo
- Placebo / Tadalafil (Active Comparator): Placebo for weeks 0-4. 10 mg/day Tadalafil: (Other Name: Cialis, Adcirca) for weeks 5-8.
  Interventions: Drug: tadalafil; Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — 50 mg/day for 4 weeks
  Other Names: Viagra; Revatio
  Arms: Placebo / Sildenafil; Sildenafil / Placebo
Drug: tadalafil — 10 mg/day for 4 weeks.
  Other Names: Cialis; Adcirca
  Arms: Placebo / Tadalafil; Tadalafil / Placebo
Drug: Placebo — Placebo 1 capsule per day for four weeks.

SUMMARY:
This study is funded by the Moody Endowment. In this project, we will investigate the potential effect of skeletal muscle nitric oxide (NO) production on skeletal muscle anabolism, muscle strength, physical function, and body composition in older individuals. Further, we will determine whether augmentation of NO-mediated signaling reduces fatigue and fatigability.

DETAILED DESCRIPTION:
The Investigators hypothesize that upregulation of skeletal muscle NO-cGMP mediated responses through phosphodiesterase (PDE) inhibition by sildenafil or tadalafil causes an acute anabolic response of skeletal muscle protein synthesis. NO is well-known to elicit vasodilation through stimulation of cGMP signaling, and NO-mediated changes in muscle perfusion may influence both skeletal muscle anabolism and perceptual fatigue. To measure skeletal muscle protein synthesis, we will infuse a stable isotope tracer of phenylalanine and measure its incorporation into skeletal muscle proteins following a dose of sildenafil, tadalafil, or placebo. The Investigators will also determine whether differences exist between men and women in response to PDE inhibition. As skeletal muscle NO-cGMP signaling has been implicated in fatigue responses, we will assess the acute effect of sildenafil and tadalafil on fatigue. Fatigue can be manifested both as a performance deficit at a local level (e.g., a reduced ability of skeletal muscle to produce power or force) as well as a subjective experience of lacking physical or mental energy. Accordingly, we will use more than one means (skeletal muscle performance, fatigue questionnaires, accelerometers) to study fatigue. The Investigators hypothesize that sildenafil or tadalafil will acutely reduce exercise-associated fatigability and skeletal muscle fatigue development

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-60 years of age
2. Ability to sign consent form (score>23 on the 30-item Mini Mental Status examination, MMSE)
3. Stable body weight for at least three months.

Exclusion Criteria:

1. Physical dependence or frailty (impairment in any of the Activities of Daily Living (ADL), history of falls (>2/year) or significant weight loss in the past year).
2. Pregnancy
3. Significant heart, liver, kidney, blood or respiratory disease.
4. Peripheral vascular disease.
5. Diabetes mellitus or other untreated endocrine disease.
6. Active cancer
7. Use of nitrates.
8. Recent (within 6 months) treatment with anabolic steroids, or corticosteroids.
9. Alcohol or drug abuse.
10. Severe depression (>5 on the 15-item Geriatric Depression Scale, GDS).
11. Cardiac abnormalities such as cardiac shunt or previously diagnosed pulmonary hypertension.
12. Systolic blood pressure <100 or>150, diastolic blood pressure <60 or 90>. This range is smaller than the acceptable range stated in the prescribing information for sildenafil/tadalafil (90/50 and <170/110).

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Sheffield-Moore, PhD, Principal Investigator — University of Texas Medical Branch, Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the community via flyers and local postings.
Pre-assignment Details: 30 subjects enrolled in this study. 6 subjects failed the screening and were withdrawn. 6 subjects chose to withdraw participation before the study began. 18 subjects began the study. 2 subjects were withdrawn during the study. 16 subjects completed the study.
Groups:
- Sildenafil, Then Placebo: Sildenafil daily (50mg/day) for weeks 0-4. Then Placebo daily for weeks 5-8.
- Tadalfil, Then Placebo: Tadalafil (10mg/day) for week 0-4. Then Placebo daily for week 5-8.
- Placebo, Then Sildenafil: Placebo daily for weeks 0-4. Then Sildenafil daily (50mg/day) for weeks 5-8.
- Placebo, Then Tadalafil: Placebo for week 0-4, then Tadalafil (10mg/day) for week 5-8.
Period: Phase 1: Week 0-4
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Started | 5 | 4 | 5 | 4
Completed | 4 | 4 | 5 | 4
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Phase 2: Week 5-8.
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Started | 4 | 4 | 5 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 30 subjects enrolled in this study. 6 subjects failed the screening and were withdrawn. 6 subjects chose to withdraw participation before the study began. 18 subjects began the study. 2 subjects were withdrawn during the study. 16 subjects completed the study.
Groups:
- Sildenafil, Then Placebo: Sildenafil (50mg/day) daily for weeks 0-4, then Placebo daily weeks 5-8.
- Tadalfil, Then Placebo: Tadalafil (10mg/day) daily for weeks 0-4, then Placebo daily for weeks 5-8.
- Placebo, Then Sildenafil: Placebo daily for weeks 0-4, then Sildenafil (50mg/day) daily for weeks 5-8.
- Placebo, Then Tadalafil: Placebo daily for weeks 0-4, then Tadalafil (10mg/day) daily for weeks 5-8.
- Total: Total of all reporting groups
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil | Total
Number analyzed (Participants) | 5 | 4 | 5 | 4 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (4.16) | 56 (1.41) | 52.4 (1.51) | 57.25 (2.99) | 54.6 (3.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 2 | 13
  Male | 1 | 0 | 2 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 5 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Skeletal Muscle Fatigue as Measured by Biodex 4 Pro After 4 Weeks of Placebo
Description: Isokinetic Fatigue Measure (knee extension) is measured on a Biodex System Pro 4 within a 75 degree range of motion. Subjects performed concentric contractions at a fixed speed of 120 degree/sec. 50 contractions were performed at 100% force, one contraction every second. Isokinetic fatigue will be measured at week 4 and week 8. Depending on grouping, the week 4 and week 8 measures may be placebo or active drug. Data will be reported as after 4 weeks of placebo or after 4 weeks of active drug. Data is presented as mean maximum force over all 50 kicks.
Time Frame: after 4 weeks of placebo
Measure: Mean (Standard Deviation); unit: Newton-Meters
Groups:
- Sildenafil, Then Placebo: 50 mg/day Sildenafil: (Other Name: Viagra, Revatio) for weeks 0-4. Placebo for weeks 5-8.
  Sildenafil: 50 mg/day for 4 weeks
  Placebo: Placebo 1 capsule per day for four weeks.
- Tadalafil, Then Placebo: 10 mg/day Tadalafil: (Other Name: Cialis, Adcirca) for weeks 0-4. Placebo for weeks 5-8.
  tadalafil: 10 mg/day for 4 weeks.
  Placebo: Placebo 1 capsule per day for four weeks.
- Placebo, Then Sildenafil: Placebo for weeks 0-4. 50 mg/day Sildenafil: (Other Name: Viagra, Revatio) for weeks 5-8.
  Sildenafil: 50 mg/day for 4 weeks
  Placebo: Placebo 1 capsule per day for four weeks.
- Placebo, Then Tadalafil: Placebo for weeks 0-4. 10 mg/day Tadalafil: (Other Name: Cialis, Adcirca) for weeks 5-8.
  tadalafil: 10 mg/day for 4 weeks.
  Placebo: Placebo 1 capsule per day for four weeks.
Arm/Group | Sildenafil, Then Placebo | Tadalafil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
Newton-Meters | 59.69 (33.71) | 42.07 (5.19) | 67.17 (26.87) | 63.24 (8.34)

2. Primary Outcome: Skeletal Muscle Fatigue as Measured by Biodex 4 Pro After 4 Weeks of Active Drug
Description: as for outcome 1
Time Frame: after 4 weeks of active drug
Measure: Mean (Standard Deviation); unit: Newton-Meters
Arm/Group | Sildenafil / Placebo | Tadalafil / Placebo | Placebo / Sildenafil | Placebo / Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
Newton-Meters | 60.90 (35.60) | 42.48 (6.30) | 62.68 (24.88) | 63.25 (15.12)

3. Primary Outcome: Exercised Induced Fatigability as Measured by Fatigue Rating Scale After 4 Weeks of Placebo
Description: The fatigue rating scale is a scale from 0 to 10 with 0 being no fatigue at all and 10 being the worst fatigue the subject can imagine. The subject is asked to rate their level of fatigue in their leg. This test was performed before and immedicately after the Biodex leg fatigue test after 4 weeks of placebo. Data is presented as change in scale from pre fatigue test to post fatigue test, with a higher score indicating a greater level of fatigue.
Time Frame: after 4 weeks of placebo
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil / Placebo | Tadalafil / Placebo | Placebo / Sildenafil | Placebo / Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
units on a scale | 4.33 (1.53) | 2.5 (0.58) | 7.0 (1.83) | 4.75 (0.96)

4. Primary Outcome: Exercised Induced Fatigability as Measured by Fatigue Rating Scale After 4 Weeks of Active Drug
Description: The fatigue rating scale is a scale from 0 to 10 with 0 being no fatigue at all and 10 being the worst fatigue the subject can imagine. The subject is asked to rate their level of fatigue in their leg. This test was performed before and immedicately after the Biodex leg fatigue test. Data is presented as change in scale from pre fatigue test to post fatigue test, with a higher score indicating a greater level of fatigue.
Time Frame: after 4 weeks of active drug
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil / Placebo | Tadalafil / Placebo | Placebo / Sildenafil | Placebo / Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
units on a scale | 4.5 (2.38) | 3.5 (1.73) | 5.25 (4.27) | 6.0 (1.83)

5. Secondary Outcome: Maximum Peak Isometric Leg Strength as Measured by Biodex Pro4 After 4 Weeks of Placebo
Description: Peak isometric strength is measured on a Biodex System 4 Pro. This test is isolated to the quadricep muscle of one leg. Isometric test is performed at 90 degrees with 5 seconds of force production for each contraction and 15 seconds of rest. 1 set of 3 contractions at 100% force performed. Isometric strength was measured at week 4 and week 8. Depending on grouping, the week 4 and week 8 measures may be placebo or active drug. Data will be reported as after 4 weeks of placebo or after 4 weeks of active drug.
Time Frame: after 4 weeks of placebo
Measure: Mean (Standard Deviation); unit: Newton-Meters
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
Newton-Meters | 145.86 (97.73) | 104.17 (23.66) | 149.14 (62.67) | 148.34 (47.26)

6. Secondary Outcome: Maximum Peak Isometric Leg Strength as Measured by Biodex Pro4 After 4 Weeks of Active Drug.
Description: as for outcome 5
Time Frame: after 4 weeks of active drug
Measure: Mean (Standard Deviation); unit: Newton-Meters
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
Newton-Meters | 140.09 (82.29) | 110.39 (21.26) | 133.81 (58.04) | 139.96 (50.47)

7. Secondary Outcome: Maximum Peak Isokinetic Leg Strength as Measured by Biodex Pro4 After 4 Weeks of Placebo.
Description: Isokinetic strength (knee extension) is measured on a Biodex System Pro 4 within a 75 degree range of motion. Subjects performed concentric contractions at a fixed speed of 120 degree/sec. 1 set of 3 contractions were performed at 100% force. Isokinetic strength will be measured at week 4 and week 8. Depending on grouping, the week 4 and week 8 measures may be placebo or active drug. Data will be reported as after 4 weeks of placebo or after 4 weeks of active drug.
Time Frame: after 4 weeks of placebo
Measure: Mean (Standard Deviation); unit: Newton-Meters
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
Newton-Meters | 105.15 (49.46) | 78.59 (10.25) | 117.71 (39.86) | 111.67 (23.43)

8. Secondary Outcome: Maximum Peak Isokinetic Leg Strength as Measured by Biodex Pro4 After 4 Weeks of Active Drug
Description: as for outcome 7
Time Frame: after 4 weeks of active drug
Measure: Mean (Standard Deviation); unit: Newton-Meters
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
Newton-Meters | 106.79 (49.69) | 79.33 (11.69) | 116.48 (37.83) | 114.75 (36.49)

9. Secondary Outcome: Lean Body Mass as Measured by Dual Energy X-ray Absorptiometry at Week 0.
Description: Lean Body Mass is calculated from a whole body scan measured on a dual energy x-ray absorptiometry.
Time Frame: week 0
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 5 | 4 | 5 | 4
kilograms | 44.60 (11.62) | 41.43 (4.72) | 49.93 (10.63) | 54.45 (14.28)

10. Secondary Outcome: Lean Body Mass as Measured by Dual Energy X-ray Absorptiometry at Week 4.
Description: Lean Body Mass is calculated from a whole body scan measured on a dual energy x-ray absorptiometry.
Time Frame: week 4
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 5 | 4
kilograms | 46.29 (14.40) | 41.02 (4.05) | 50.61 (10.67) | 54.85 (14.71)

11. Secondary Outcome: Lean Body Mass as Measured by Dual Energy X-ray Absorptiometry at Week 8.
Description: Lean Body Mass is calculated from a whole body scan measured on a dual energy x-ray absorptiometry.
Time Frame: week 8
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
kilograms | 46.22 (14.68) | 40.76 (4.38) | 52.09 (10.03) | 55.10 (14.42)

12. Secondary Outcome: Fat Mass as Measured by Dual Energy X-ray Absorptiometry at Week 0.
Description: Fat Mass is calculated from a whole body scan measured on a dual energy x-ray absorptiometry.
Time Frame: week 0
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 5 | 4 | 5 | 4
kilograms | 32.35 (11.40) | 37.21 (6.81) | 32.72 (5.92) | 32.10 (6.90)

13. Secondary Outcome: Fat Mass as Measured by Dual Energy X-ray Absorptiometry at Week 4.
Description: Fat Mass is calculated from a whole body scan measured on a dual energy x-ray absorptiometry.
Time Frame: week 4
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 5 | 4
kilograms | 33.16 (12.42) | 37.12 (6.35) | 32.30 (5.55) | 32.47 (7.08)

14. Secondary Outcome: Fat Mass as Measured by Dual Energy X-ray Absorptiometry at Week 8.
Description: Fat Mass is calculated from a whole body scan measured on a dual energy x-ray absorptiometry.
Time Frame: week 8
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
kilograms | 33.60 (12.51) | 37.02 (6.21) | 32.40 (5.83) | 32.79 (7.12)

15. Secondary Outcome: Walking Distance at 100% Effort as Measured by Walking Test After 4 Weeks of Placebo
Description: Walking performance will be assessed during 2 minutes of walking in long corridor hallways. Subjects will be asked to walk at 100% effort (as quickly as they can safely walk without running) for 2 minutes. Distance traveled for the 2 minutes will be recorded. The walking test will be completed at week 4 and week 8. Depending on grouping, the week 4 and week 8 measures may be placebo or active drug. Data will be reported as after 4 weeks of placebo or after 4 weeks of active drug.
Time Frame: after 4 weeks of placebo
Population: 1 subject did not complete the walking test
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 3 | 4 | 4 | 4
meters | 203.82 (30.51) | 189.79 (38.12) | 198.41 (14.04) | 202.80 (37.84)

16. Secondary Outcome: Walking Distance at 100% Effort as Measured by Walking Test After 4 Weeks of Active Drug
Description: as for outcome 15
Time Frame: after 4 weeks of active drug
Population: 1 subject did not complete the walking test.
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 3 | 4 | 4 | 4
meter | 197.01 (32.72) | 178.56 (17.84) | 200.19 (13.99) | 203.46 (31.11)

17. Secondary Outcome: Perceptual Fatigue as Measured by Multidimensional Fatigue Symptom Inventory - Short Form Total Score at Week 0
Description: Fatigue symptoms will be measured using the 30-item Multidimensional Fatigue Symptom Inventory - Short Form, a validated measure that yields one overall score of total fatigue calculated using five sub scales (general, physical, emotional, mental, vigor). With the exception of the vigor sub scale, higher scores indicate greater fatigue. Total fatigue score is calculated by summing the sub categories (general, physical, emotional and mental) and subtracting vigor. Total scores range from -24 to 96, with a higher score indicating more fatigue.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
scores on a scale | 9.66 (19.55) | -7.5 (5.45) | -8 (3.61) | -3.75 (9.54)

18. Secondary Outcome: Perceptual Fatigue as Measured by Multidimensional Fatigue Symptom Inventory - Short Form Total Score at Week 4
Description: as for outcome 17
Time Frame: week 4
Population: 1 subject did not complete the week 4 MFSI questionnaire
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 3 | 4 | 4
scores on a scale | 6.33 (26.08) | -3.33 (10.97) | -6.33 (2.31) | -3.5 (12.66)

19. Secondary Outcome: Perceptual Fatigue as Measured by Multidimensional Fatigue Symptom Inventory - Short Form Total Score at Week 8
Description: as for outcome 17
Time Frame: week 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
scores on a scale | 9.67 (19.09) | 3.25 (27.54) | -9.67 (6.81) | -9.25 (1.26)

20. Other Pre Specified Outcome: Hemoglobin Level at Week 0
Description: Hemoglobin was measured by University of Texas Medical Branch Clinical Laboratory. Normal ranges are 11.6 - 15.0 g/dL.
Time Frame: week 0
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
g/dL | 13.42 (0.97) | 12.78 (0.71) | 12.4 (0.53) | 13.05 (0.90)

21. Other Pre Specified Outcome: Hemoglobin Level Measured at Week 4
Description: Hemoglobin was measured by University of Texas Medical Branch Clinical Laboratory. Normal ranges are 11.6 - 15.0 g/dL.
Time Frame: week 4
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
g/dL | 13.05 (0.49) | 12.03 (0.43) | 12.6 (0.37) | 13.2 (0.47)

22. Other Pre Specified Outcome: Hemoglobin Level Measured at Week 8
Description: Hemoglobin was measured by University of Texas Medical Branch Clinical Laboratory. Normal ranges are 11.6 - 15.0 g/dL.
Time Frame: week 8
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
g/dL | 13.55 (0.35) | 11.97 (0.76) | 12.5 (0.08) | 12.95 (1.17)

23. Other Pre Specified Outcome: Hematocrit Level Measured at Week 0
Description: Hematocrit was measured by University of Texas Medical Branch Clinical Laboratory. Normal ranges are 35.7 - 45.2%.
Time Frame: week 0
Measure: Mean (Standard Deviation); unit: percent of red blood cells
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
percent of red blood cells | 39.53 (2.16) | 38.55 (1.42) | 37.25 (2.07) | 31.88 (13.09)

24. Other Pre Specified Outcome: Hematocrit Level Was Measured at 4 Weeks
Description: Hematocrit was measured by University of Texas Medical Branch Clinical Laboratory. Normal ranges are 35.7 - 45.2%.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percent of red blood cells
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
percent of red blood cells | 39.08 (0.84) | 37.38 (0.82) | 38.13 (0.77) | 39.1 (1.81)

25. Other Pre Specified Outcome: Hematocrit Level Measured at Week 8
Description: Hematocrit was measured by University of Texas Medical Branch Clinical Laboratory. Normal ranges are 35.7 - 45.2%.
Time Frame: week 8
Measure: Mean (Standard Deviation); unit: percent of red blood cells
Arm/Group | Sildenafil, Then Placebo | Tadalfil, Then Placebo | Placebo, Then Sildenafil | Placebo, Then Tadalafil
Number analyzed (Participants) | 4 | 4 | 4 | 4
percent of red blood cells | 40.38 (0.44) | 36.6 (1.94) | 38.1 (1.19) | 38.4 (3.24)

ADVERSE EVENTS:
Groups:
- Sildenafil: Sildenafil (50mg/day) daily for 4 weeks.
- Tadalfil: Tadalafil (10mg/day) daily for 4 weeks.
- Placebo: Placebo daily for week 4 weeks.
Arm/Group | Sildenafil | Tadalfil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/18
Other Adverse Events (participants affected / at risk) | 2/10 | 0/8 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=10) | Tadalfil (N=8) | Placebo (N=18)
Redness at site of muscle biopsy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (General disorders) | 1 (1) | 0 (0) | 0 (0) — Syncope following administration of Sildenafil 50mg.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No